CLINICAL TRIAL: NCT00284843
Title: The Epidemiology of Group A Streptococcal Infections in Fiji (Fiji GrASP) Part 1: The Prevalence of Rheumatic Heart Disease, Pyoderma and Scabies in School Children in Fiji
Brief Title: Prevalence of RHD, Pyoderma and Scabies in Children in Fiji
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0118
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2007-10

CONDITIONS: Streptococcus Group A
Keywords: Streptococcus, Fiji, pyoderma, scabies, rheumatic disease
MeSH Terms: conditions — Pyoderma; Scabies; Rheumatic Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to estimate the number of cases of rheumatic heart disease, pyoderma, and scabies in school age children in Fiji. In addition the study will describe the features of rheumatic heart disease, pyoderma, and scabies in these children. Study participants will include 5200 primary school children, ages 5-14, from 21 primary schools in the Central Division of Fiji. These children will be examined for pyoderma, scabies, and the doctor will listen to their heart with a stethoscope. Any child that has a heart murmur detected will have their heart looked at through an echocardiogram test (uses sound waves to create a picture of how the heart is working). Any child that is found to have rheumatic heart disease will be referred to a pediatric cardiologist for further evaluation. Participants will be involved in the study for about 2 days.

DETAILED DESCRIPTION:
This study is the first of 5 studies (including DMID protocols 05-0081, 05-0082, 05-0117, and 06-0081) in a larger project aimed at evaluating the epidemiology of infections caused by the group A streptococcus (GAS) in Fiji - this larger project is called the Fiji Group A Streptococcal Project (Fiji GrASP). Fiji GrASP is in turn part of a larger program aimed at progression of a novel GAS vaccine - this program is the project entitled "Global GAS Vaccine Based On The M-Protein". The three broad aims of the Fiji GrASP epidemiologic studies are to: establish the burden of disease of GAS infections in Fiji; describe the molecular epidemiology of GAS isolates in Fiji; and establish natural immunologic correlates of protection of a J8 vaccine if they exist. The Fiji GrASP epidemiologic studies are important for vaccine clinical trials in that they will gain a clear picture of the burden of GAS disease, develop ongoing surveillance and clinical endpoints for vaccine trials, collect isolates of GAS in Fiji, investigate immune correlates of vaccine protection, and prepare the existing clinical trial site for trials of the J-8 based vaccine. The primary objectives of this study are to estimate the prevalence of rheumatic heart disease (RHD) in primary school aged children in Fiji and to estimate the prevalence of pyoderma in these children. Secondary objectives are to: estimate the prevalence of scabies in primary school aged children in Fiji; describe the clinical and echocardiographic features of RHD in these children; and describe the clinical features of pyoderma and scabies in these children. Approximately 5,200 primary school children, 5-14 years of age, from 21 primary schools in the Central Division of Fiji will participate in this study. They will be examined for pyoderma and scabies, and they will have a standard auscultation by a pediatrician. Any child with a murmur will have a screening echocardiogram of the mitral and aortic valves. If abnormality of these valves is identified or if another pathology is suspected, the child will be referred to a pediatric cardiologist for full echocardiogram. The primary endpoints of the study will be to determine the prevalence of echocardiogram confirmed rheumatic heart disease and to determine the prevalence of pyoderma assessed using a standardized tool. The secondary endpoints will be to determine: prevalence of scabies assessed using a standardized tool; prerevalence of heart failure or signs of ventricular enlargement in children with echocardiographically-confirmed RHD; distribution and severity of valvular lesions in children with echocardiographically-confirmed RHD; prevalence of severe pyoderma and body distribution (upper vs lower) of lesions; and prevalence of scabies, severe scabies and body distribution (upper vs lower) of scabies lesions.

ELIGIBILITY:
Inclusion Criteria:

All children between the ages of 5 to 14 years of age within the schools identified will be eligible to participate in the study and provide informed consent.

Exclusion Criteria:

None identified

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5200
Dates: Start 2006-01; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Locations (1):
- Colonial War Memorial Hospital, Suva, Fiji